CLINICAL TRIAL: NCT03379090
Title: Using In-depth Interviews to Examine Neighborhood Influence on Parenting Practices Regarding Youth Outdoor Play and Physical Activity.
Brief Title: Neighborhood Influence on Parenting Practices Regarding Youth Outdoor Play
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Maura Kepper, Postdoctoral Fellow, Pennington Biomedical Research Center
Other Study IDs: 2017-017-PBRC; 1F32HD093282-01 (NIH)
Record Dates: First submitted 2017-12-12; First posted 2017-12-20 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Physical Activity; Adolescent Behavior; Parenting
MeSH Terms: conditions — Motor Activity; Adolescent Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parental constraint of outdoor play may be fueling unhealthy emotional and physical development in today's children and adolescents. Time spent outdoors is a key determinant of unstructured play and overall physical activity levels, both of which are crucial to optimal development in youth. Modern barriers - such as crime, poor social ties among neighbors, and unsafe physical environments - constrain parental practices and reduce opportunities for outdoor play in children and youth. Low levels of perceived collective efficacy, a measure of perceived neighborhood cohesion and the collective capacity to solve neighborhood problems, has been proposed as a social environmental factor that constrains outdoor play by parents either attempting to avoid potentially dangerous situations or using defensive behavior by upgrading security measures. Moreover, incivilities in the neighborhood physical environment (e.g. litter, graffiti, blighted property) may influence parents' perceived collective efficacy. Consequently, a child's ability to achieve the recommended minimum of 60 minutes of daily physical activity may be limited by a complex interaction between neighborhood social and physical environmental factors and the extent to which parents respond by constraining offspring outdoor play. The central hypothesis of this research is that modifiable factors in the neighborhood social and physical environment result in parental constraint of offspring outdoor play, which reduces overall physical activity during critical years of development. This research will use qualitative methods to generate a comprehensive understanding of how and which environmental factors play a crucial role in parental constraint of outdoor play and promote low levels of within-neighborhood physical activity. This ancillary study will recruit 32 parents/guardians of participants from the parent study, Translational Investigation of Growth and Everyday Routines in Kids (TIGER Kids) Study (USDA 3092-51000-056-04A), to participate in in-depth interviews. My ultimate goal is to use knowledge gained from this ancillary study to generate community-based interventions that will target neighborhood factors to successfully reduce parental constraints on outdoor play.

ELIGIBILITY:
Inclusion Criteria:

-Child completed baseline measures (Y0) for the parent study, TIGER Kids Study (USDA 3092-51000-056-04A).

Exclusion Criteria:

* Child did not complete baseline measures (Y0) of the TIGER Kids Study.
* Did not report a home address at the baseline (Y0) TIGER Kids study visit.
* Unwilling or unable to participate in an in-depth interview.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 32 parents/guardians of participants from the TIGER Kids parent study will be recruited for this study. All parents/guardians will be recruited after their child has completed the baseline (Y0) TIGER Kids study visit.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Perceptions of how the social environment influences parenting practices related to outdoor play and youth's physical activity. | One time-point, 1 hour in-depth interview
  Indepth interviews will be used to measure parental perceptions of how the social environment in which they live influences their parenting decisions regarding their child's outdoor play.

CONTACTS AND LOCATIONS:
Overall Officials: Maura Kepper, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share IPD. Qualitative data may be difficult to prepare to ensure privacy of the participant. Furthermore, we do not see the benefit of sharing IPD from this study as qualitative data cannot be easily reanalyzed to validate study findings, combined with other datasets, and has a high risk of being analyzed using invalid/non-rigorous methods.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT03379090/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT03379090/ICF_001.pdf